Title: Noninvasive NAVA Versus NIPPV in Low Birthweight Premature Infants

NCT #: NCT03137225

Document approval date: 09/08/2016

Document Type: Protocol and Statistical Analysis Plan

Date: Thursday, September 08, 2016 12:49:46 PM

View: SF - Study Identification

Print Close

# Study Identification

1. \* Select the Principal Investigator:

Henry Rozycki

2. \* Study Title:

ID: HM20005575

Noninvasive NAVA Versus NIPPV in Low Birthweight Premature Infants

- 3. \* Is this a student or trainee project in which activities will be carried out by that individual under your supervision:
  - YesNo
- 4. Select any associated VCU IRB protocols:

ID PI

There are no items to display

Select all individuals who are permitted to edit the IRB protocol and should be copied on communications (study staff will be entered later). These individuals will be referred to as protocol editors:

| Last Name | First Name | E-Mail | Phone | Mobile |
|-----------|------------|--------|-------|--------|

ID: HM20005575

View: SF - Student/Trainee Investigator Contact



ID: HM20005575

View: SF - Research Determination

#### Research Determination

1. \* Select one of the following that applies to the project:

- Research Project or Clinical Investigation

  Exception from Informed Consent for Planned Emergency Research

  Humanitarian Use of Device for Treatment or Diagnosis

  Humanitarian Use of Device for Clinical Investigation

  Emergency Use of Investigational Drug, Biologic or Device

  Treatment Use (Expanded Access to Investigational Product for Treatment Use)

  Center or Institute Adminstrative Grant Review
- ID: HM20005575

View: SF - Federal Regulations

# Federal Regulations

- 1. \* Is this a Clinical Trial:
  - Yes
  - O No
- 2. Is this an Applicable Clinical Trial that must be registered and reported to clinicaltrials.gov:
  - No
- 3. \* Is this a FDA regulated study:
  - Yes
  - No
- 4. \* Is this study supported by the Department of Defense (DoD):
  - No.
  - No
- 5. \* Check if any of the following funding sources apply to this research:

None of the above

ID: HM20005575 View: SF - Personnel

## Personnel

1. \* Indicate all VCU/VCUHS personnel, including the PI, who will be engaged in this study:



Identify all non-VCU personnel who will be engaged in this study AND who DO NOT have IRB approval for this study from their own institution.

Name Roles Roles - Other Responsibilities - Qualifications Qualifications COI Investigator

There are no items to display

3. CV/Biosketch: (required for PI, Medically/Psychologically Responsible Investigators and Student/Trainee Investigators)

ID: HM20005575

View: SF - Conflict of Interest

## Conflict of Interest

- 1. \* To the best of your knowledge, do you (as PI) or any other engaged individual hold a financial conflict of interest related to this study?
  - Yes
  - No
- 2. If Yes, provide:
  - Name(s) of the engaged conflicted individual(s)
  - Brief description of the financial conflict of interests
- 3. \* Describe any potential non-financial conflicts of interest for members of the research team that could impact the conduct of the study (if None, please state "None"):
- 4. Describe any institutional conflict of interest with this research that you or any member of the research team may be aware of:

  None

ID: HM20005575

View: SF - Communication Plan for Research Team

#### Communication Plan for Research Team

1. \* Describe the process that will be used to ensure that all persons at all involved sites assisting with the research are adequately informed about the protocol and their research related duties and functions: Investigators will brief and inform clinical personnel of study design by poster in break room, email and personal interactions before first enrollment; however, clinical personnel will be not be performing any research related duties. Members of the research team will meet after each subject to review protocol, data acquisition and to go over any problems identified.

# IRB Panel Setup

1. \* To which IRB is this study being submitted for review:

| VCU IRB |
|-----------------------------------------------------|
| Western IRB |
| NCI Central IRB |
| Other IRB (Request to Defer to Another Institution) |

ID: HM20005575

View: SF - Review Setup

# Review Setup

1. \* Does this study involve greater than minimal risk:

Yes No

2. \* Review Type Requested: (subject to IRB approval)

| Full Board |
|------------|
| Expedited |
| Exempt |

ID: HM20005575

View: SF - Research Description

## Research Description

1. \* Describe the study hypothesis and/or research questions. Use lay language whenever possible.

We hypothesize that in very low birth weight infants who require respiratory support via noninvasive ventilation, that synchronizing the ventilator breath with the baby's breath using neurally adjusted ventilatory assist (NAVA) will reduce the number and/or severity of apnea/bradycardia/desaturation episodes compared to nasal intermittent positive pressure ventilation (NIPPV).

2. \* Describe the study's specific aims or goals. Use lay language whenever possible.

The specific goal is to measure the number and severity of cessation of breath/low heart rate/low blood oxygen level events (ie, apnea/bradycardia/desaturation events) in a 4 hour period while receiving one of the two types of non-invasive ventilation modes (either NIPPV or NAVA) currently used in very low birthweight infants.

3. \* Describe the study's background and significance, including citations, or upload a citation list in document upload. Use lay language whenever possible.
Very low birthweight (VLBW) premature infants in the NICU frequently require respiratory support for prolonged periods of time. Invasive

Very low birthweight (VLBW) premature infants in the NICU frequently require respiratory support for prolonged periods of time. Invasive mechanical ventilation (which requires intubating the baby with a tube to provide breaths) can lead to ventilator-induced lung injury. Because of this, noninvasive respiratory support has become increasingly popular, as this form of ventilation has been shown to reduce the incidence of permanent lung injury. (1)

There are several methods to provide non-invasive support. The gentlest is continual flow of air and oxygen via nasal cannula. However, premature infants often develop apnea, either becasue the signals from their immature brain are not yet sufficient or because the muscles in the back of their throat do not get enough nerve signals to maintain sufficient opening. As a result, babies on nasal cannula often develop clinical apnea/bradycardia/desaturations. Before putting these babies back on invasive ventilation, clinicians often try to provide the baby with machine breaths while still on non-invasive ventilation. This method is called nasal intermittent positive pressure ventilation and studies have demonstrated that this method reduces the need for re-intubation in VLBW infants (1) and reduces the rate of apneic events.

A newer method of non-invasive breathing support that has been FDA approved and used in VLBW infants, synchronizes the machine generated breath with the patient's own breath. Neurally adjusted ventilatory assist (NAVA) does this by replacing the standard nasogastric tube with a nasograstric tube that has sensors which detect the baby's natural diaphragm activity, which signal the ventilator to breath in synchronization with the baby. Studies have shown that the efficacy of nasal ventilation is significantly enhanced when the machine breath is synchronized with the patient breath (2). Synchronization also reduces diaphragmatic dysfunction (3). It can improve gas delivery, reduce work of breathing, and make patients demonstrably more comfortable (4).

Neurally Adjusted Ventilatory Assist (NAVA) is a mode of partial support. NAVA can be used both in intubated patients (invasive NAVA) as well as in extubated patients who require noninvasive positive pressure ventilation (noninvasive NAVA) (5). Invasive NAVA has been shown to deliver equivalent ventilation while requiring lower peak inspiratory pressure, as well as reduced respiratory muscle load, compared to conventional pressure support ventilation.

Currently, the choice of using NIPPV or NAVA is at the clinician's discretion. Both are regularly and frequently used in the VCU Health System's NICU. There are no studies that have examined whether NAVA triggered synchronized ventilation is more effective than non-synchronized NIPPV. In addition, there is limited data on the synchronicity and mechanics of non-invasive NAVA in VLBW infants. Information comparing clinical and lung mechanical outcomes between NIPPV and NIV NAVA would significantly benefit VLBW care providers and, consequently, their patients in getting the best evidenced-based therapy.

- 1. Tang S, Zhao J, Shen J, Hu Z, Shi Y. Nasal intermittent positive pressure ventilation versus nasal continuous positive airway pressure in neonates: a systematic review and meta-analysis. Indian Pediatr. 2013 Apr;50(4):371-6.
- 2. Gizzi C, Montecchia F, Panetta V, Castellano C, Mariani C, Campelli M, Papoff P, Moretti C, Agostino R. Is synchronised NIPPV more effective than NIPPV and NCPAP in treating apnoea of prematurity (AOP)? A randomised cross-over trial. Arch Dis Child Fetal Neonatal Ed. 2015 Jan; 100(1):F17-23.
- 3. Petrof B, Jaber S, Matecki S. Ventilator-induced diaphragmatic dysfunction. Current opinion in critical care 2010; 16(1): 19-25
- 4. Stein H, Firestone K. Application of neurally adjusted ventilatory assist in neonates. Seminars in Fetal and Neonatal Medicine 2014; 19(1): 60-69.
- 5. Moerer O, Beck J, Brander L, Costa R, Quintel M, Slutsky AS, et al. Subject-ventilator synchrony during neural versus pneumatically triggered non-invasive

helmet ventilation. Intensive Care Med 2008: 34:1615-23

4. \* Briefly describe the study design, including all interventions or interactions with research participants and access to identifiable data. Use lay language whenever possible.

#### a. Subjects

Subjects: VLBW (< 1501 grams birthweight) infants in the VCU Health System NICU who are receiving either NPPV or non-inasive NAVA therapy as ordered by their clinical providers. Investigators are clinicians who work in the NICU and will therefore be able to identify eliminate subjects

NAVA and NIPPV are different modes for the way non-invasive ventilation breaths are triggered. Both utilize the same delivery system, ventilator, cannula, etc. In NIPPV, the ventilator breaths are triggered by time, i.e. the ventilator sends a breath to match the prescribed rate like one every 3 seconds for a rate of 20 breaths per minute, no matter whether the patient is inhaling or exhaling. In NAVA, the normal feeding tube is replaced by a special tube that has a sensor located around where the diaphragm surrounds the esophagus. The sensor picks up the electrical signal of the diaphragm muscle contracting, and this mark of the beginning of inhalation is used to trigger a machine breath, so the machine and the patient are coordinated. Aside from the catheter connection, all other procedures are the same. b). Randomization - the order of modes will be assigned based on a random number table using a 5 block design to match the DSMB reporting needs. c) The change from one mode to the next involves activating a switch on the ventilator. There are no procedures that need to be done to the subject. They will remain in their current environment, connected to all the routine and study-related monitoring equipment. d) During the study, which involves both modes, the subjects will be monitored as routine by the staff, as well as one of the study faculty (Rozycki or Moores). In the event that one of us needs to step away briefly, an attending neonatologist and a neonatal fellow are on site in the NICU

As part of routine care, infants on either mode have a nasograstric tube in place. Those subjects who are receiving NIPPV will have their nasogastric tubes replaced by a NAVA nasograstric tube. The subject will then be randomized to one of the two modes (NIPPV or non-invasive NAVA). After a one hour stabilization period, during which small adjustments to the non-inasive settings can be made to clinically optimize the settings, the study will begin. A Nellcor pulse oximeter probe will be placed on an extremity to provide a continuous non-invasive downloadable measure of saturation (blood oxygen level) and heart rate. Data from the ventilator will be downloaded in real-time to a laptop. These data will be recorded for 4 hours continuously. After that, the ventiliator will be switched to the other mode (NIPPV to NAVA or NIPPV), at the same PEEP and respiratory rate. Again, one hour will be allowed to adjust the ventilator settings. Data will then be collected for 4 hours on the second ventilation mode. At that time, the clinician will be informed if either mode was significantly better and the clinician will decide which mode the patient will return to. We will not know which mode is better until the data are analyzed in aggregate. We're concerned about safety perspective where the subject is on Mode A as chosen by the clinician, and we find that during the time they are on Mode A, they have far more events than when we have them on Mode B. This would be valuable information, since the choice of NPIIV vs. NAVA is currently not clearly indicated. To address this, we will provide the clinician with the results that are available at the time of the study. This will be number of events that are routinely measured clinically, i.e. events that cause alarms such as apnea or bradycardia or desaturations outside the clinical limits. These are objective measures that the clinician can incorporate into their decision making if they so choose.

Data to be collected will include heart rate, saturations from the pulse oximeter, and respiratory rate, expired tidal volume, peak pressure and synchronization from the ventilator.

Clinical data will include: birthweight, gestational age, age at study (days of life) and pre-study ventilator settings, Data will be kept in a secure HIPAA compliant database and only study investigators will have access to it.

Analysis: The simultaneous recordings will be scored for: a) Apnea ( cessation of breath resulting in no airflow for > 20 seconds or for > 5 seconds if accompanied by bradycardia [HR < 100 bpm] or desaturation [Oximetry < 85%]) b) Bradycardia (hr < 100 bpm for > 5 seconds) c) Desaturation (< 85% for > 5 seconds) d) Synchronicity, measured as average triggering and cycling-off delays for each modality, and total wasted patient respiratory efforts for each modality.

Primary outcome: The number of isolated apneas, bradycardias and desaturations and the number of combined events will be compared by mode of ventilation.

Secondary outcome: a) Synchronicity from the ventilator at the time of an event. This will be analyzed to determine whether asynchronicity is related to increased number of events during the study. b) Overall asynchronicity counts will be determined by ventilator data that can be uploaded and analyzed with software supplied by the manufacturer. c) average mean airway pressure and peak inspiratory pressures required in each mode of ventilation.

There are no well-characterized tools to measure premature infant 'comfort'. There are semi-subjective pain scores that the nursing staff use but we are more likely to have irritation or discomfort from the probe. Thus, this will be an ongoing assessment of a) the infant's state - quiet sleep, quiet awake, agitated, restless, etc. b) new onset tachycardia or tachypnea coincident with applying the probes. c) facial grimaces that are different than baseline as assessed by the nurse caring for the patient

The threshold for an adverse event will be dependent on the baseline level. If the baseline rate is, say, 4-6 events an hour, a 25% increase is 1 event, which is within the patient's variance. On the other hand, in one having no events, just one event is a 100% increase. We have 2 criteria - 1) An event that requires intervention with breathing support such as with more breaths or a bag and mask, 2) an increase from baseline of at least 4-5 events/hr. from baseline

5. Upload any supporting tables or documents:

ID: HM20005575 View: SF - Study Activities

#### Study Activities

| 1. * Select which study type | best describes the majority | of the study. Your response | will help determine which | ı IRB panel should |
|---|---|---|---|---|
| review this. | | | | |

| • | Bio-Medical |
|---|---|
| 0 | Qualitative - Social/Behavioral/Education (SBE) |
| 0 | Quantitative - SBE |
| 0 | Mixed Method - SBE |
| 0 | Mixed Method - Biomedical |
| * Th | is study will involve (check all that apply): |
| | procedures such as surveys, interviews, field studies, focus groups, educational tests, deception, psycho-physiological testing, any other similar data collection |
| | secondary data analysis: procedures such as analysis of information collected for non-research purposes (includes both retrospective and prospectively collected information), or analysis of data previously collected for a prior research study |

drugs, devices, experimental interventions, biohazards, radiation, other medical or surgical procedures

ID: HM20005575 View: SF - Bio-Med Project Details

# Bio-Med Project Details

#### 1. \* Select all details that apply:

| | Drugs, Biologics, | Supplements, and/or Other Co | mpounds | | |
|---|---|---|---|---|---|
| | | | <u> </u> | | |
| | Placebo | | | | |
| | Washout Period | | | | |
| • | Device Evaluation | on | | | |
| | Bio-Hazards, Oth | er Toxins, Recombinant DNA/0 | Gene Transfer | | |
| | Radiation Exposure and/or Scans involving radiation (PET, MRA) | | | | |
| | Stem Cells | | | | |
| | Expanded Access - Treatment Use of an Investigational Product | | | | |
| | Other Medical or | Surgical Procedures | | | |
| <b>✓</b> | Protected Health | n Information (PHI) | | | |
| HM200 | 005575 | View: SF - Bio-Med | l Device Evalua | ation Details | |
| | | evice Evaluation evice evaluation this study w | | 6 | |
| • | Marketed Medica | al Device (including 510k dev | vice) | | |
| | Investigational Me | edical Device | | | |
| | New Use for Mark | keted Medical Device | | | |
| | Other Devices | | | | |
| 2. * Li | ist devices this stu | udy will involve: | | | |
| De | evice | Manufacturer | IDE | IDE Holder | Doc |
| Ser | rvo-i Ventilator | Maquet | N/A | Not Required | Servo-i (0.01) |
| Ser | rvo-i NAVA | Maquet | N/A | Not Required | NAVA brochure(0.01) |
| | number: Study I Commi | Protocol including IDE numb<br>unication from the FDA with<br>eld by the sponsor, upload at | er<br>verification of | the IDE | ring documents for verification of the ID |
| | number: Study I Comm If the IDE is he (required if IN) Sponse Commi | eld by a sponsor-investigator Protocol including IDE numb unication from the FDA with eld by the sponsor, upload at D held by sponsor): or protocol unication from the sponsor v unication from the FDA verification | verification of<br>t least one of the<br>verifying the III | the IDE<br>the following docum<br>DE number<br>umber | ents for verification of the IDE number |
| | number: Study I Comm If the IDE is he (required if IN) Sponse Commi | eld by a sponsor-investigator Protocol including IDE numb unication from the FDA with eld by the sponsor, upload at D held by sponsor): or protocol unication from the sponsor v | verification of<br>t least one of the<br>verifying the III | the IDE<br>the following docum<br>DE number<br>umber | ents for verification of the IDE number |
| НМ200 | number: Study I Commi If the IDE is he (required if IN) Sponse Commi Commi | eld by a sponsor-investigator Protocol including IDE numb unication from the FDA with eld by the sponsor, upload at D held by sponsor): or protocol unication from the sponsor w unication from the FDA verify un approved device, upload d | verification of<br>t least one of the<br>verifying the III | the IDE the following docum The number umber and the approved us | ents for verification of the IDE number |
| | number: Study I Commi If the IDE is h (required if IN) Sponse Commi Commi | Protocol including IDE numb<br>unication from the FDA with<br>eld by the sponsor, upload at<br>D held by sponsor):<br>or protocol<br>unication from the sponsor v<br>unication from the FDA verify<br>in approved device, upload d | verification of<br>t least one of the<br>verifying the II<br>ying the IDE not<br>documentation | the IDE the following docum The number umber and the approved us | ents for verification of the IDE number |
| | number: Study I Commi If the IDE is he (required if IN) Sponse Commi Commi | Protocol including IDE numb<br>unication from the FDA with<br>eld by the sponsor, upload at<br>D held by sponsor):<br>or protocol<br>unication from the sponsor v<br>unication from the FDA verify<br>in approved device, upload d | verification of<br>t least one of the<br>verifying the II<br>ying the IDE not<br>documentation | the IDE the following docum The number umber and the approved us | ents for verification of the IDE number |
| ata | number: Study I Commi If the IDE is h (required if IN) Sponse Commi Commi | Protocol including IDE numb unication from the FDA with eld by the sponsor, upload at D held by sponsor): or protocol unication from the sponsor vunication from the FDA verify in approved device, upload diview: SF- | verification of<br>t least one of the<br>verifying the II<br>ying the IDE not<br>documentation | the IDE the following docum The number umber and the approved us | ents for verification of the IDE number |
| ata | number: Study I Commi If the IDE is he (required if IN) Sponse Commi Commi Formation Commi | Protocol including IDE numb<br>unication from the FDA with<br>eld by the sponsor, upload at<br>D held by sponsor):<br>or protocol<br>unication from the sponsor v<br>unication from the FDA verifi<br>un approved device, upload d<br>View: SF - | verification of<br>t least one of the<br>verifying the II<br>ying the IDE not<br>documentation | the IDE the following docum The number umber and the approved us | ents for verification of the IDE number |
| ata<br>1. * se | number: Study I Commi If the IDE is he (required if IN) Sponse Commi Commi If evaluating a | Protocol including IDE numb unication from the FDA with eld by the sponsor, upload at D held by sponsor): or protocol unication from the sponsor vunication from the FDA verify in approved device, upload diview: SF-IDE Tails IDE Tails In the study: | verification of<br>t least one of the<br>verifying the II<br>ying the IDE not<br>documentation | the IDE the following docum The number umber and the approved us | ents for verification of the IDE number |
| ata | number: Study I Commi If the IDE is he (required if IN) Sponse Commi Commi Commi Commi Commi Commi Specimen/Biologi Protected Health | Protocol including IDE numb<br>unication from the FDA with<br>eld by the sponsor, upload at<br>D held by sponsor):<br>or protocol<br>unication from the sponsor v<br>unication from the FDA verifi<br>un approved device, upload d<br>View: SF - | verification of<br>t least one of the<br>verifying the II<br>ying the IDE not<br>documentation | the IDE the following docum The number umber and the approved us | ents for verification of the IDE number |
| ata<br>1. * se | number: Study I Commi If the IDE is he (required if IN) Sponse Commi Commi Gommi If evaluating a | Protocol including IDE numb unication from the FDA with eld by the sponsor, upload at D held by sponsor): or protocol unication from the sponsor vunication from the FDA verifies approved device, upload diview: SF-IDE TAILS in the study: c Sample Collection Information (PHI) | verification of<br>t least one of the<br>verifying the III<br>ying the IDE in<br>documentation<br>- Data Collection | the IDE the following docum The following docum The number The infinite approved us The provided in the provid | ents for verification of the IDE number |
| ata<br>1. * se | number: Study I Commi If the IDE is he (required if IN) Sponse Commi Commi Commi Fevaluating a | Protocol including IDE numb unication from the FDA with eld by the sponsor, upload at D held by sponsor): or protocol unication from the sponsor v unication from the FDA verify in approved device, upload d View: SF | verification of<br>t least one of the<br>verifying the III<br>ying the IDE in<br>documentation<br>- Data Collection | the IDE the following docum The following docum The number The infinite approved us The provided in the provid | ents for verification of the IDE number |
| ata<br>1. * se | number: Study I Commi If the IDE is he (required if IN) Sponse Commi Commi Commi Fevaluating a | Protocol including IDE numb unication from the FDA with eld by the sponsor, upload at D held by sponsor): or protocol unication from the sponsor vunication from the FDA verifies an approved device, upload diview: SF-IDETAILS in the study: In Cample Collection Information (PHI) | verification of the least one of the lea | the IDE the following docum DE number umber of the approved us on Details | ents for verification of the IDE number |
| ata<br>1.*se | number: Study I Commi If the IDE is he (required if IN) Sponse Commi Commi Commi Fevaluating a Co5575 Collection Specimen/Biologi Protected Health Audio/Video Existing Data or S Use of Internet for Registries/Reposi | Protocol including IDE numb unication from the FDA with eld by the sponsor, upload at D held by sponsor): or protocol unication from the sponsor v unication from the FDA verify in approved device, upload d View: SF - Details in the study: ic Sample Collection in Information (PHI) Specimens Not From a Registry r Data Collection itories (Includes Accessing, Co | verification of the least one of the lea | the IDE the following docum DE number umber of the approved us on Details | ents for verification of the IDE number |
| ata 1. * \$6 | number: Study I Commi If the IDE is he (required if IN) Sponse Commi Comm | Protocol including IDE numb unication from the FDA with eld by the sponsor, upload at D held by sponsor): or protocol unication from the sponsor vunication from the FDA verifies approved device, upload diview: SF-ID Details in the study: In Cample Collection Information (PHI) Specimens Not From a Registry r Data Collection intories (Includes Accessing, Come | verification of the least one of the lea | the IDE the following docum DE number umber of the approved us on Details | ents for verification of the IDE number |
| ata 1. * \$6 | number: Study I Commi If the IDE is he (required if IN) Sponse Commi Commi Commi Fevaluating a Co5575 Collection elect all involved i Specimen/Biologi Protected Health Audio/Video Existing Data or S Use of Internet for Registries/Reposi None of the Abov elect all identifiers an if the data will e | Protocol including IDE numb unication from the FDA with eld by the sponsor, upload at D held by sponsor): or protocol unication from the sponsor v unication from the FDA verifi un approved device, upload of View: SF - Details In the study: C Sample Collection Information (PHI) Specimens Not From a Registry IT Data Collection itories (Includes Accessing, Co | verification of the least one of the lea | the IDE the following docum DE number umber of the approved us on Details | ents for verification of the IDE number |
| ata 1. * \$6 | number: Study I Commi If the IDE is he (required if IN) Sponse Commi C | Protocol including IDE numb unication from the FDA with eld by the sponsor, upload at D held by sponsor): or protocol unication from the sponsor wunication from the FDA verify an approved device, upload of View: SF - Details In the study: In Specimens Not From a Registry or Data Collection interior (Includes Accessing, Collection interior (Includes Accessing)) | verification of the least one of the lea | the IDE the following docum DE number umber of the approved us on Details | ents for verification of the IDE number |
| ata 1. * \$6 | number: Study I Commi If the IDE is he (required if IN) Sponse Commi Commi Commi Fevaluating a costs of Internet for Registries/Reposition of the Abovelect all identifiers in the data will e Names Geographic Local | Protocol including IDE numb unication from the FDA with eld by the sponsor, upload at D held by sponsor): or protocol unication from the sponsor vunication from the FDA verify in approved device, upload diview: SF-IDE Tails in the study: In Cample Collection Information (PHI) Specimens Not From a Registry r Data Collection itories (Includes Accessing, Collection in Information (PHI)) State of the study in the study in the study in the study: In Cample Collection in the specimens in the study in the stud | verification of the least one of the lea | the IDE the following docum DE number umber of the approved us on Details | ents for verification of the IDE number |
| ata 1. * \$6 | number: Study I Commi If the IDE is he (required if IN) Sponse Commi C | Protocol including IDE numb unication from the FDA with eld by the sponsor, upload at D held by sponsor): or protocol unication from the sponsor wunication from the FDA verify in approved device, upload diview: SF - Details in the study: or Sample Collection in Information (PHI) Specimens Not From a Registry or Data Collection itories (Includes Accessing, Collection itories (Includes Accessing, Collection itories Selow State Level umbers | verification of the least one of the lea | the IDE the following docum DE number umber of the approved us on Details | ents for verification of the IDE number |
| ata 1. * \$6 | number: Study I Commi If the IDE is he (required if IN) Sponse Commi C | Protocol including IDE numb unication from the FDA with eld by the sponsor, upload at D held by sponsor): or protocol unication from the sponsor vunication from the FDA verify in approved device, upload diview: SF-IDE Tails in the study: In Cample Collection Information (PHI) Specimens Not From a Registry r Data Collection itories (Includes Accessing, Collection in Information (PHI)) State of the study in the study in the study in the study: In Cample Collection in the specimens in the study in the stud | verification of the least one of the lea | the IDE the following docum DE number umber of the approved us on Details | ents for verification of the IDE number |

| | Facsimile Numbers | |
|---|---|---|
| | E-mail Addresses | |
| • | Medical Record Numbers | |
| • | Device Identifiers | |
| | Biometric Identifiers | |
| | Web URLs | |
| | IP Addresses | |
| | Account Numbers | |
| | Health Plan Numbers | |
| | Full Face Photos or Comparable Images | |
| | License/Certification Numbers | |
| | Vehicle ID Numbers | |
| | Other Unique Identifier | |
| | No Identifiers | |
| | Employee V# | |
| part | Vill participants be able to withdraw their data (participate:<br>) Yes<br>) No | per, electronic, or specimens) from the study if they no longer wish to |
| part<br>• | rticipate: Yes | |
| part in the second sec | rticipate: Yes No ves above, describe how participants will be able 005575 | |
| part Description The description PAA Description Des | rticipate: Yes No No res above, describe how participants will be able 005575 A rescribe the protected health information that will RN, birth dates, date of study. The only data that are redications while on study, ventilator mode and settings rescribe the source(s) of the protected health info 8.U's electronic medical record system cxplain how the PHI collected or used in this resear e above mentioned data will be needed to evaluate the scriptors of a neonatal research population (birth-weig | to withdraw their data: View: SF - HIPAA be obtained or used in this research: needed from the EMR are: gestational age, birth-weight, age at study, s at time of study, gender and Apgar scores and head ultrasound results. remation: arch is the minimum necessary to accomplish this research: ne role of maturity on the outcomes. These variables are either standard clinically, gestational age, gender, Apgar Scores) to inform any reader of an imple is representative of the relevant population, or ones that can influence the |
| part Description The description PAA Description Des | res above, describe how participants will be able to 2005575 A rescribe the protected health information that will seem that date of study. The only data that are redications while on study, ventilator mode and settings the scribe the source(s) of the protected health inforture electronic medical record system explain how the PHI collected or used in this research above mentioned data will be needed to evaluate the scriptors of a neonatal research population (birth-weig gregated data publication about whether the study satcome variable (medications, ventilator history, evider the select all pathways this research will employ to us | to withdraw their data: View: SF - HIPAA be obtained or used in this research: needed from the EMR are: gestational age, birth-weight, age at study, s at time of study, gender and Apgar scores and head ultrasound results. remation: arch is the minimum necessary to accomplish this research: ne role of maturity on the outcomes. These variables are either standard clinically, gestational age, gender, Apgar Scores) to inform any reader of an imple is representative of the relevant population, or ones that can influence the |
| part Description The description PAA Description Des | rticipate: Yes No res above, describe how participants will be able 1005575 A rescribe the protected health information that will 1005575 Rescribe the protected health information that are redications while on study, ventilator mode and settings rescribe the source(s) of the protected health informations while on study, ventilator mode and settings rescribe the source(s) of the protected health informations will be record to system of the protected health information has been supported by the protected or used in this researce above mentioned data will be needed to evaluate the scriptors of a neonatal research population (birth-weig gregated data publication about whether the study satcome variable (medications, ventilator history, evider relect all pathways this research will employ to us | to withdraw their data: View: SF - HIPAA be obtained or used in this research: needed from the EMR are: gestational age, birth-weight, age at study, s at time of study, gender and Apgar scores and head ultrasound results. remation: arch is the minimum necessary to accomplish this research: ne role of maturity on the outcomes. These variables are either standard clinically, gestational age, gender, Apgar Scores) to inform any reader of an imple is representative of the relevant population, or ones that can influence the |
| part Description The description PAA Description Des | res above, describe how participants will be able to the protected health information that will be able to the protected health information that will be able to the protected health information that are reductions while on study, ventilator mode and settings describe the source(s) of the protected health information while on study, ventilator mode and settings the source(s) of the protected health information will be needed to evaluate the scriptors of a neonatal research population (birth-weig gregated data publication about whether the study accome variable (medications, ventilator history, evider telect all pathways this research will employ to us to be ledentified Data Limited Data Set | to withdraw their data: View: SF - HIPAA be obtained or used in this research: needed from the EMR are: gestational age, birth-weight, age at study, s at time of study, gender and Apgar scores and head ultrasound results. remation: arch is the minimum necessary to accomplish this research: ne role of maturity on the outcomes. These variables are either standard clinically, gestational age, gender, Apgar Scores) to inform any reader of an imple is representative of the relevant population, or ones that can influence the |
| part Description The description PAA Description Des | res above, describe how participants will be able to the protected health information that will RN, birth dates, date of study. The only data that are redications while on study, ventilator mode and settings the scribe the source(s) of the protected health information while on study, ventilator mode and settings the scribe the source(s) of the protected health information has been solved to the protected of the protected health information will be needed to evaluate the scriptors of a neonatal research population (birth-weig pregated data publication about whether the study satisfactories are provided to the study satisfactories are provided to the study satisfactories and pathways this research will employ to use the left of the protected and pathways this research will employ to use the protected and pathways the protected and pathw | to withdraw their data: View: SF - HIPAA be obtained or used in this research: needed from the EMR are: gestational age, birth-weight, age at study, s at time of study, gender and Apgar scores and head ultrasound results. remation: arch is the minimum necessary to accomplish this research: ne role of maturity on the outcomes. These variables are either standard clinically, gestational age, gender, Apgar Scores) to inform any reader of an imple is representative of the relevant population, or ones that can influence the |
| part PA | res above, describe how participants will be able to the protected health information that will be able to the protected health information that will be able to the protected health information that are restricted in the protected health are restricted by the protected health information while on study, ventilator mode and settings to the source(s) of the protected health information how the PHI collected or used in this researe above mentioned data will be needed to evaluate the scriptors of a neonatal research population (birth-weig gregated data publication about whether the study accome variable (medications, ventilator history, evider telect all pathways this research will employ to us be-Identified Data Limited Data Set Waiver of Authorization Partial Waiver of Authorization | be obtained or used in this research: needed from the EMR are: gestational age, birth-weight, age at study, s at time of study, gender and Apgar scores and head ultrasound results. rmation: arch is the minimum necessary to accomplish this research: ne role of maturity on the outcomes. These variables are either standard clinicaght, gestational age, gender, Apgar Scores) to inform any reader of an imple is representative of the relevant population, or ones that can influence the core of brain bleeds) se or access PHI: |
| part Description The description PAA Description Des | res above, describe how participants will be able to the protected health information that will RN, birth dates, date of study. The only data that are redications while on study, ventilator mode and settings the scribe the source(s) of the protected health information while on study, ventilator mode and settings the scribe the source(s) of the protected health information has been solved to the protected of the protected health information will be needed to evaluate the scriptors of a neonatal research population (birth-weig pregated data publication about whether the study satisfactories are provided to the study satisfactories are provided to the study satisfactories and pathways this research will employ to use the left of the protected and pathways this research will employ to use the protected and pathways the protected and pathw | be obtained or used in this research: needed from the EMR are: gestational age, birth-weight, age at study, s at time of study, gender and Apgar scores and head ultrasound results. rmation: arch is the minimum necessary to accomplish this research: ne role of maturity on the outcomes. These variables are either standard clinica ght, gestational age, gender, Apgar Scores) to inform any reader of an imple is representative of the relevant population, or ones that can influence the core of brain bleeds) se or access PHI: |

# Data Confidentiality and Storage

1. \* Confidentiality refers to the way private, identifiable information about a participant or defined community is maintained and shared. Describe all of the precautions that will be used to maintain the confidentiality of identifiable information, samples or

Subjects will have a study number unique to the subject. The key linking the study number to the patient will be kept in a separate comouter file stored in a password protected computer and file. All other data will be stored in VCU RedCap files.

The data on the laptop is non-identifiable. It will consist of real-time data from the ventilator and apnea monitor, without any identifiers. It will be analyzed for events, without identifiers. Only the event numbers (number and duration of apneas, bradycardias, etc. and synchronicity) will be linked to the subject when stored in VCU Redcap files. The signed consent form will be stored in a locked filing cabinet in a locked office in the VCU Children's Pavilion.

2. \* Who will have access to study data:

- 3.  $^{\circ}$  If applicable, describe the process for assigning codes to the data including : how codes will be assigned

  - whether there will be a key linking identifiable information to the data
     where the key will be stored
     who will have access to the key

- when the key will be destroyed
Each subject will get a study number (1, 2, 3, etc) as they are identified/consented to the study. The code will be kept separately as above and access limited to study investigators. The key code will be destroyed upon completion of tfe study and analysis. The key linking the study number to the patient will be kept in a separate computer file stored in a password protected computer and file. Only the 4 investigators named in this study (Moores, Xu, Sirota and Rozycki) will have access to the key.

4. \* Will the sponsor or investigator obtain a certificate of confidentiality for this study:

| No. CoC will not be Obt | ained |
|---|---|
| No - CoC will not be Obt Yes - CoC has been Obta | |
| Yes - CoC Request is Pen | • |
| Yes - Plan to Submit CoC | Request |
| 5. If the Certificate of Confiden | tiality has been obtained by the PI, upload it here: |
| 6. * What will happen to the res | search records when the research has been completed: |
| Stored indefinitely with ide | entifiers removed |
| Stored indefinitely with ide | entifiers attached |
| <ul> <li>Destroyed at the end of<br/>Policy and/or sponsor re</li> </ul> | study once the minimum time required for data retention has been met per VCU Data Retention stanting requirements |
| Destroyed when notified b | by sponsor but not less than the minimum time required for data retention per VCU Data Retention Policy |
| Other | |
| 7. If Other, explain: | |
| | lentifiers attached", explain why identifiers are necessary: |
| HM20005575 | View: SF - Types of Sites |
| pes of Sites | |
| • | ng accurately describes this study: |
| Not Multicenter Study | |
| Multicenter Study - VCU L | ead |
| Multicenter Study - Non-V | CU Lead |
| 2. * Select all sites where study | y interventions or interactions will occur and/or identifiable data will be held: |
| <b>VCU Site</b> | |
| Non-VCU Site (VCU Inve | stigators are conducting/overseeing the conduct of the study) |
| 3. * Is there a community parts Yes No | ner in this research study: |
| HM20005575 | View: SF - VCU Site Details |
| CU Site Details | |
| 1. * Select all VCU sites that wi | Il be utilized in this study: |
| Clinical Research Service | se Unit (CRSU) |
| Massey Cancer Center | · '' |
| ✓ VCU Health System | |
| VCU Qatar | |
| Site - NICU on CCH6 | |
| HM20005575 | View: SF - VCU Health System |
| CU Health Syster | n |
| 1. * The PI has reviewed and as policy: Yes | grees to comply with the Conduct of Clinical Research in VCU Health System Patient Care Areas |
| ○ No | |

2. \* Explain how you will notify and obtain support from patient care providers in the units where the study will be conducted: Investigators will brief and inform clinical personnel of study design by poster in break room, email and personal interactions before first enrollment.

ID: HM20005575 View: SF - Study Funding

| 1 | | ave you applied for funding:<br>Yes |
|---|---|---|
| | | No |
| 2 | $\subset$ | o, is this study already funded:<br>) Yes<br>) No |
| о. н | พวกก | 005575 View: SF - Study Population |
| J. 11 | VIZUC | 10075 Hell: el. Clady i spalate. |
| Stu | ıdy | Population |
| 1 | . <b>* P</b> ı<br>15 | rovide the total number of participants you expect to enroll in this study under the VCU IRB: |
| 2 | . If ti | nis is a multi-Center Project, what is the total anticipated number of subjects across all sites: |
| 3 | | rovide justification for the sample size:<br>mple Size |
| | 0.0 | sed on published data, monitored events occur at an average frequency of 9.2 over a 4-hour period. The degree of variability is not own but assuming an SD of 50%, a sample size of 10 subjects would have an 0.8 power for a 50% reduction in events at an alpha of 5. A similar study to ours comparing NIPPV and flow-synchronized NIPPV (2) had 19 participants and achieved statistically significant arences between the two modalities. Based on this, we are anticipating a need for 15 subjects |
| 4 | 1. <<br>2. F | st the study inclusion criteria:<br>: 1501 grams (VLBW infant)<br>Patient must be receiving daily caffeine therapy for apnea<br>On non-invasive ventitation, either NIPPV or non-invasive NAVA |
| 5 | | st the study exclusion criteria: |
| | for | No concerns for acute sepsis (i.e., blood cultures, if drawn, have been negative 48 hours, and no active signs/symptoms of sepsis). |
| | 3. N | No history of meningitis or seizures No signs of increased intracranial pressure, including bulging fontanelle, presence of ventricular shunt device, or ventriculomegaly by st recent ultrasound. |
| | 4, F | screem unrasound. Presence of Grade III or IV intraventricular hemorrhage to cyanotic heart defects or clinically significant congenital heart disease. Will allow PDA, PFO, and mild to moderate ASD/VSD as |
| | det | to cyanotic hear to defects of children's significant congenital heart disease. Will allow PDA, PPO, and fillid to moderate ASD/VSD as ermined by pediatric cardiology. John-English speaking legal representatives (parents) |
| 6 | | heck all participant groups that are likely to be involved in this study. If it is possible that a regulated vulnerable population |
| | | ildren, pregnant women, prisoners) COULD BE involved in the study, be sure to check them: |
| | | Healthy Valuntaers |
| | | Healthy Volunteers |
| | <b>V</b> | Children |
| | | Emancipated Minors |
| | _ | Pregnant Women |
| | = | Fetuses, Neonates, Fetal Material or In-Vitro Fertilization |
| | | Decisionally Impaired Adults |
| | | When cancer is integral to the research - cancer Patients, Family Members, Healthcare Providers or Prevention |
| | | VCU Health System Patients |
| | | Non-VCU Patients |
| | | VCU/VCUHS Students or Trainees |
| | | VCU/VCUHS Employees |
| | | Individuals with Limited English Proficiency |
| | | Active Military Personnel |
| | | When researching in a K-12 environment - populations Within School Districts or Other Learning Environments |
| 7 | gro<br>The<br>or a | ou are either targeting, or excluding, a particular segment of the population / community, provide a description of the up/organization/community and provide a rationale: e decreased ability to explain the technical aspects of the study to LEP parents through either medically-approved translation service medically-certified informed consent form in other languages makes it difficult for these parents to be fully informed to make a ision in the best interests of their child. |
| 8 | . * S | elect the age range(s) of the participants who may be involved in this study: |
| | 4 | <1 Year |
| | | 1 - 6 Years |
| | | 7 - 12 Years |
| | | 1 - 14 IVAIS |
| | | 12 17 Voors |
| | | 13 - 17 Years |
| | | 18 - 20 Years |

ID: HM20005575 View: SF - Children

| | _ | | | |
|---|---|---|---|---|
| | | 45<br>CFF<br>46.4 | child | arch involving no greater than minimal risk to children, with adequate provisions for soliciting the assent of the ren and permission of their parents or guardians, as set forth in Sec. 46.408 |
| | 1 | 45<br>CFR<br>46.4 | t parti | arch involving greater than minimal risk but presenting the prospect of direct benefit to individual cipants |
| | | 45<br>CFF<br>46.4 | gene | arch involving greater than minimal risk and no prospect of direct benefit to individual participants, but likely to yield ralizable knowledge about the participant s disorder or condition |
| | | 45<br>CFF<br>46.4 | R affec | arch not otherwise approvable which presents an opportunity to understand, prevent or alleviate a serious problem ting the health or welfare of children. (Research in this category must be reviewed and approved by the Secretary experiment of Health & Human Services) |
| 2. | $\subset$ | /ill thi | s study | involve participants who could be wards of the state: |
| 3. | | | e how | children will be assented to participate in the study: |
| 4 | | | | nis study is recruiting newborn infants only |
| 4. | Par<br>with | rents o | of stable<br>an-term | /ou plan to obtain permission of parents or guardians:<br>infants receiving non-invasive ventilation will be approached in their private single patient NICU rooms and presented<br>information about the study. They will be given a copy of the consent form, all of their questions will be answered and<br>opportunity to take the information home to review. |
| : HN | 1200 | 00557 | 5 | View: SF - Children: Direct Benefit [45 CFR 46.405] |
| hi | ldı | ren | : Dir | ect Benefit [45 CFR 46.405] |
| 1. | | | | how the risk is justified by the anticipated benefit to participants: |
| | ma<br>wat<br>brie | y be b<br>tches | etter. He<br>for clinic<br>od of tim | s of non-invasive ventilation are currently approved and used in the US and in the VCU NICU, it is not known which<br>ence, there is a possibilty that one mode may be inferior to the other. Currently, a clinician picks one mode and then<br>al signs to determine if they picked the right one. By participating in this study, the subject gets exposed to both in a<br>e, and the efficacy and superiority of one over the other can be assessed. In normal care, this side by side assessmen |
| 2. | | | | how the relation of the anticipated benefit to the risk is at least as favorable to the participants as that ailable alternative approaches: |
| | The | e alter | native a | proach is to not participate. Study participants will be far more intensely monitored for how the ventilation mode is<br>-participants. Non-participants depend on nursing observation (a nurse may have 1-2 other patients) and historic data |
| | bet | ter ab | le to ass | Participants will have an investigator watching their respiratory status continuously for four hours on each mode, so be<br>ess which one is better for the subject. This information will be shared with the clinical team who may use it to<br>a better mode of non-invasive ventilation for that patient. |
| | | 00557 | | View: SF - Pregnant Women, Fetuses, Neonates and Post-Delivery Material |
| re | gr | nan<br><sub>heck</sub> | t Wo | omen, Fetuses, Neonates and Post-Delivery Material e following categories that apply to this research: |
| re | gr | nan<br><sub>heck</sub> | all of th | omen, Fetuses, Neonates and Post-Delivery Material |
| re | gr | 1 <b>a</b> n<br>heck | all of th | omen, Fetuses, Neonates and Post-Delivery Material e following categories that apply to this research: 204 Research involving pregnant women or fetuses. Research involving neonates of uncertain viability. |
| re | gr | 45 C<br>45 C<br>46.2<br>(b) | all of the | omen, Fetuses, Neonates and Post-Delivery Material e following categories that apply to this research: 204 Research involving pregnant women or fetuses. Research involving neonates of uncertain viability. |
| re | gr | 45 C<br>45 C<br>46.2<br>(b)<br>45 C<br>46.2<br>(c) | all of th<br>CFR 46.2<br>CFR 205(a) an | omen, Fetuses, Neonates and Post-Delivery Material e following categories that apply to this research: 204 Research involving pregnant women or fetuses. Research involving neonates of uncertain viability. |
| re | gr | 45 C<br>45 C<br>46.2<br>(b)<br>45 C<br>46.2<br>(c) | of Wo | omen, Fetuses, Neonates and Post-Delivery Material e following categories that apply to this research: 204 Research involving pregnant women or fetuses. Research involving neonates of uncertain viability. Research involving nonviable neonates |
| re | gr | 45 C<br>45 C<br>46.2<br>(b)<br>45 C<br>46.2<br>(c) | all of the<br>CFR 46.2<br>CFR 05(a) and<br>CFR 05(a) and<br>CFR 05(d) | omen, Fetuses, Neonates and Post-Delivery Material e following categories that apply to this research: 204 Research involving pregnant women or fetuses. Research involving neonates of uncertain viability. Research involving nonviable neonates Research involving viable neonates. |
| re | gr<br>*c | 45 C<br>45 C<br>46.2<br>(b)<br>45 C<br>46.2<br>(c) | t Wo<br>all of th<br>EFR 46.2<br>EFR 05(a) al<br>EFR 05(d) al<br>EFR 05(d) | omen, Fetuses, Neonates and Post-Delivery Material of following categories that apply to this research: Out Research involving pregnant women or fetuses. Research involving neonates of uncertain viability. Research involving nonviable neonates Research involving viable neonates. Out Research involving, after delivery, the placenta, the dead fetus, or fetal material. |
| 1. | gr<br>* c | 45 C<br>45 C<br>45 C<br>46 C<br>(b)<br>45 C<br>46 C<br>45 C | t We will be seen the control of the | omen, Fetuses, Neonates and Post-Delivery Material of following categories that apply to this research: Out Research involving pregnant women or fetuses. Research involving neonates of uncertain viability. Research involving nonviable neonates Research involving viable neonates. Out Research involving, after delivery, the placenta, the dead fetus, or fetal material. Out Research involving, after delivery, the placenta and opportunity to understand, prevent, or alleviate a serious problem affecting the health or welfare of pregnant women, fetuses, or neonates. |
| 1. | gr<br>* c | 45 C 46.2 (b) 45 C 46.2 (c) 45 C 45 C 45 C 45 C | t Wo | omen, Fetuses, Neonates and Post-Delivery Material of following categories that apply to this research: Out Research involving pregnant women or fetuses. Research involving neonates of uncertain viability. Research involving nonviable neonates Research involving viable neonates. Out Research involving, after delivery, the placenta, the dead fetus, or fetal material. Out Research involving, after delivery, the placenta, the dead fetus, or neonates and provent, or alleviate a serious problem affecting the health or welfare of pregnant women, fetuses, or neonates. View: SF - Neonates: Viable [45 CFR 46.205d] |
| 1. | gr<br>* c | 45 C 46.2 (b) 45 C 46.2 (c) 45 C 45 C 45 C 45 C 45 C 45 C 45 C 45 | t Wo | omen, Fetuses, Neonates and Post-Delivery Material of following categories that apply to this research: Out Research involving pregnant women or fetuses. Research involving neonates of uncertain viability. Research involving nonviable neonates Research involving viable neonates. Out Research involving, after delivery, the placenta, the dead fetus, or fetal material. Out Research not otherwise approvable which presents an opportunity to understand, prevent, or alleviate a serious problem affecting the health or welfare of pregnant women, fetuses, or neonates. View: SF - Neonates: Viable [45 CFR 46.205d] is collected on a neonate (newborn, after delivery) that is VIABLE, the regulations for special protections for |
| 1.<br>ec | gr<br>* c | 45 C 46.2 (b) 45 C 46.2 (c) 45 C 45 C 45 C 45 C 45 C 45 C 45 C 45 | t Wo | omen, Fetuses, Neonates and Post-Delivery Material e following categories that apply to this research: 204 Research involving pregnant women or fetuses. Research involving neonates of uncertain viability. Research involving nonviable neonates of uncertain viability. Research involving viable neonates. 206 Research involving, after delivery, the placenta, the dead fetus, or fetal material. 207 Research not otherwise approvable which presents an opportunity to understand, prevent, or alleviate a serious problem affecting the health or welfare of pregnant women, fetuses, or neonates. View: SF - Neonates: Viable [45 CFR 46.205d] is collected on a neonate (newborn, after delivery) that is VIABLE, the regulations for special protections for Subpart D). Therefore, in addition to selecting Viable neonates here, Children must be selected in Study is collected on pregnant women, or the viability of the neonate is questioned, other sections may apply. |
| 1.<br>ec | gr<br>* c | 45 C 46.2 (b) 45 C 46.2 (c) 45 C 45 C 45 C 45 C 45 C 45 C 45 C 45 | t Wo | omen, Fetuses, Neonates and Post-Delivery Material a following categories that apply to this research: 204 Research involving pregnant women or fetuses. Research involving neonates of uncertain viability. Research involving nonviable neonates Research involving viable neonates 206 Research involving, after delivery, the placenta, the dead fetus, or fetal material. 207 Research not otherwise approvable which presents an opportunity to understand, prevent, or alleviate a serious problem affecting the health or welfare of pregnant women, fetuses, or neonates. View: SF - Neonates: Viable [45 CFR 46.205d] is collected on a neonate (newborn, after delivery) that is VIABLE, the regulations for special protections for Subpart D). Therefore, in addition to selecting Viable neonates here, Children must be selected in Study |
| re 1. eu | gr<br>* c | 45 C 46.2 (b) 45 C 46.2 (c) 45 C 46.2 (c) 45 C 46.2 (c) 45 C 45 C 45 C 45 C 45 C 45 C 45 C 45 | t Wo | omen, Fetuses, Neonates and Post-Delivery Material e following categories that apply to this research: 204 Research involving pregnant women or fetuses. Research involving neonates of uncertain viability. Research involving nonviable neonates of uncertain viability. Research involving viable neonates. 206 Research involving, after delivery, the placenta, the dead fetus, or fetal material. 207 Research not otherwise approvable which presents an opportunity to understand, prevent, or alleviate a serious problem affecting the health or welfare of pregnant women, fetuses, or neonates. View: SF - Neonates: Viable [45 CFR 46.205d] is collected on a neonate (newborn, after delivery) that is VIABLE, the regulations for special protections for Subpart D). Therefore, in addition to selecting Viable neonates here, Children must be selected in Study is collected on pregnant women, or the viability of the neonate is questioned, other sections may apply. |
| re 1. eu | gr<br>* c | 45 C 45 C 46.2 (b) 45 C 46.2 (c) 45 C 45 C 45 C 45 C 45 C 45 C 45 C 45 | t Wo<br>all of th<br>EFR 46.2<br>EFR 05(a) all<br>EFR 46.3<br>EFR 46.3<br>EFR 46.3<br>EFR 46.3<br>EFR 46.3<br>EFR 46.3 | omen, Fetuses, Neonates and Post-Delivery Material of following categories that apply to this research: 104 Research involving pregnant women or fetuses. Research involving neonates of uncertain viability. Research involving nonviable neonates Research involving viable neonates 105 Research involving, after delivery, the placenta, the dead fetus, or fetal material. 106 Research involving, after delivery, the placenta, the dead fetus, or fetal material. 107 Research not otherwise approvable which presents an opportunity to understand, prevent, or alleviate a serious problem affecting the health or welfare of pregnant women, fetuses, or neonates. View: SF - Neonates: Viable [45 CFR 46.205d] Is collected on a neonate (newborn, after delivery) that is VIABLE, the regulations for special protections for subpart D). Therefore, in addition to selecting Viable neonates here, Children must be selected in Study is collected on pregnant women, or the viability of the neonate is questioned, other sections may apply. View: SF - Potential Subject Identification and Recruitment beject Identification and Recruitment ruitment methods that may be used: |
| re 1. eu | gr<br>* c | 45 C 46.2 (b) 45 C 46.2 (c) 45 C 46.2 (c) 45 C 45 C 45 C 45 C 45 C 45 C 45 C 45 | t Wo | omen, Fetuses, Neonates and Post-Delivery Material of following categories that apply to this research: 104 Research involving pregnant women or fetuses. Research involving neonates of uncertain viability. Research involving nonviable neonates of a Research involving nonviable neonates. 105 Research involving viable neonates. 106 Research involving, after delivery, the placenta, the dead fetus, or fetal material. 107 Research not otherwise approvable which presents an opportunity to understand, prevent, or alleviate a serious problem affecting the health or welfare of pregnant women, fetuses, or neonates. 108 View: SF - Neonates: Viable [45 CFR 46.205d] 109 Is collected on a neonate (newborn, after delivery) that is VIABLE, the regulations for special protections for Subpart D). Therefore, in addition to selecting Viable neonates here, Children must be selected in Study is collected on pregnant women, or the viability of the neonate is questioned, other sections may apply. 105 View: SF - Potential Subject Identification and Recruitment beject Identification and Recruitment ruitment methods that may be used: |
| re 1. eu | gr<br>* c | 45 C 45 C 45 C 46.2 (b) 45 C 46.2 (c) 45 C 45 C 45 C 45 C 45 C 45 C 45 C 45 | t Wo all of the EFR 46.2 EFR 46.2 EFR 05(a) all EFR 05(d) EFR 46.2 EFR 46.3 EFR 46.3 EFR 46.3 EFR 46.3 EFR 46.3 EFR 46.3 EFR 46.3 | omen, Fetuses, Neonates and Post-Delivery Material of following categories that apply to this research: 104 Research involving pregnant women or fetuses. Research involving neonates of uncertain viability. Research involving nonviable neonates of a Research involving nonviable neonates. 105 Research involving viable neonates. 106 Research involving, after delivery, the placenta, the dead fetus, or fetal material. 107 Research not otherwise approvable which presents an opportunity to understand, prevent, or alleviate a serious problem affecting the health or welfare of pregnant women, fetuses, or neonates. 108 View: SF - Neonates: Viable [45 CFR 46.205d] 109 Is collected on a neonate (newborn, after delivery) that is VIABLE, the regulations for special protections for Subpart D). Therefore, in addition to selecting Viable neonates here, Children must be selected in Study is collected on pregnant women, or the viability of the neonate is questioned, other sections may apply. 105 View: SF - Potential Subject Identification and Recruitment beject Identification and Recruitment ruitment methods that may be used: |

| ļ | | |
|---|---|---|
| | 1 | Direct Contact |
| ĺ | | Psychology Research |
| ļ | | Participant Pool (SONA) |
| I | | VCU TelegRAM announcement |
| Ī | | Word of Mouth |
| Ī | | Other |
| | | her, please describe:<br>ect the methods used to obtain names and contact information for potential subjects: |
| Ī | 1 | Pre-Existing Relationship with Participants |
| Ī | | Selected from Pre-Existing VCU Records |
| Ī | | Selected from Pre-Existing Non-VCU Records |
| Ī | | Selected from Publicly Available Records |
| Ī | | Referred by Health Care Provider or Other Health Professional |
| Ī | | Recruited from Database or Registry |
| | | Identified through Community Based Organization (Schools, Church Groups, etc.) |
| - | | Self Referred (Flyer/Ad) |
| - | | Other |
| 4. I | f Ot | ner, please describe: |
| 7. U<br>F8. *<br>B8. * | When part work Family Description of Ye | |
| 1. *<br>P<br>ii<br>-<br>- | viola<br>parti<br>nfor<br>Desc<br>ide<br>rec<br>scr | vacy is an individual ♦s right to control how others view, record, or obtain information about them. When privacy is ted it can involve such things as being asked personal questions in a public setting; being publicly identified as having a cular characteristic or diagnosis; being photographed, videotaped or observed without consent; or disclosing personal mation. This is the how participants' privacy will be protected during: ntification, ruitment, seening, |
| 1. *<br>v<br>p<br>ii<br>-<br>-<br>- | Priviola<br>parti<br>nfor<br>Desc<br>ide<br>rec<br>scr<br>the<br>cor<br>dat | vacy is an individual♦s right to control how others view, record, or obtain information about them. When privacy is ted it can involve such things as being asked personal questions in a public setting; being publicly identified as having a cular characteristic or diagnosis; being photographed, videotaped or observed without consent; or disclosing personal mation. seribe how participants' privacy will be protected during: how par |
| 1. * P P P P P P P P P P P P P P P P P P | Priviola<br>parti<br>nfor<br>Desc<br>ide<br>rec<br>scr<br>the<br>cor<br>dat | vacy is an individual sright to control how others view, record, or obtain information about them. When privacy is ted it can involve such things as being asked personal questions in a public setting; being publicly identified as having a cular characteristic or diagnosis; being photographed, videotaped or observed without consent; or disclosing personal mation. seribe how participants' privacy will be protected during: https://doi.org/10.000/10.0000/10.00000000000000000000 |
| . * v Fii C T b C | Priviolation of the local control of the local cont | vacy is an individual ⊕s right to control how others view, record, or obtain information about them. When privacy is ted it can involve such things as being asked personal questions in a public setting; being publicly identified as having a cular characteristic or diagnosis; being photographed, videotaped or observed without consent; or disclosing personal mation. wribe how participants' privacy will be protected during: ntification, ruitment, sening, consent process, duct of the study, and a dissemination: VICU is a single bed room design. All work including obtaining consent, and performing the study will be done in the private single from. will only be reported in aggregate, not by individuals. No data will be linked to any information that could identify the subject |
| 1. * v F F F F F F F F F F F F F F F F F F | Priviola<br>parti<br>infor<br>Desc<br>ide<br>rec<br>scr<br>the<br>cor<br>dat | vacy is an individual ⊕s right to control how others view, record, or obtain information about them. When privacy is ted it can involve such things as being asked personal questions in a public setting; being publicly identified as having a cular characteristic or diagnosis; being photographed, videotaped or observed without consent; or disclosing personal mation. wribe how participants' privacy will be protected during: ntification, ruitment, sening, consent process, duct of the study, and a dissemination: NICU is a single bed room design. All work including obtaining consent, and performing the study will be done in the private single com. |
| 1. * P | Priviolation for the control of the | vacy is an individual stript to control how others view, record, or obtain information about them. When privacy is ted it can involve such things as being asked personal questions in a public setting; being publicly identified as having a cular characteristic or diagnosis; being photographed, videotaped or observed without consent; or disclosing personal mation. wribe how participants' privacy will be protected during: ntification, ruitment, seening, consent process, iduct of the study, and a dissemination: NICU is a single bed room design. All work including obtaining consent, and performing the study will be done in the private single com. will only be reported in aggregate, not by individuals. No data will be linked to any information that could identify the subject **To Participants** **To Participants** |
| 1. * P | Priviolation for the correction of the correctio | racy is an individual stright to control how others view, record, or obtain information about them. When privacy is ted it can involve such things as being asked personal questions in a public setting; being publicly identified as having a cular characteristic or diagnosis; being photographed, videotaped or observed without consent; or disclosing personal mation. seribe how participants' privacy will be protected during: hittication, ruitment, seening, consent process, dute to fithe study, and a dissemination: NICU is a single bed room design. All work including obtaining consent, and performing the study will be done in the private single room. will only be reported in aggregate, not by individuals. No data will be linked to any information that could identify the subject View: SF - Costs to Participants to Participants ct all categories of costs that participants or their insurance companies will be responsible for: |
| 1. * v p iii | Priviolation for Privio | racy is an individual stript to control how others view, record, or obtain information about them. When privacy is ted it can involve such things as being asked personal questions in a public setting; being publicly identified as having a cular characteristic or diagnosis; being photographed, videotaped or observed without consent; or disclosing personal mation. Pribe how participants' privacy will be protected during: hitfication, ruitment, sening, consent process, duct of the study, and a dissemination: NICU is a single bed room design. All work including obtaining consent, and performing the study will be done in the private single com. will only be reported in aggregate, not by individuals. No data will be linked to any information that could identify the subject **To Participants** **To Participants** **To Participants will have no costs associated with this study** |
| 1. * v p iii | Priviolation for ide ide received the correct the corr | racy is an individual so right to control how others view, record, or obtain information about them. When privacy is ted it can involve such things as being asked personal questions in a public setting; being publicly identified as having a cular characteristic or diagnosis; being photographed, videotaped or observed without consent; or disclosing personal mation. Trible how participants' privacy will be protected during: ntification, ruitment, beening, consent process, iduct of the study, and a dissemination: NICU is a single bed room design. All work including obtaining consent, and performing the study will be done in the private single oom. Will only be reported in aggregate, not by individuals. No data will be linked to any information that could identify the subject To Participants To Participants To Participants will have no costs associated with this study Study related procedures that would be done under standard of care |
| 1. * P | Privilation of the latest of t | racy is an individual so right to control how others view, record, or obtain information about them. When privacy is ted it can involve such things as being asked personal questions in a public setting; being publicly identified as having a cular characteristic or diagnosis; being photographed, videotaped or observed without consent; or disclosing personal mation. In the how participants' privacy will be protected during: intification, ruitment, seening, consent process, iduct of the study, and a dissemination: INCU is a single bed room design. All work including obtaining consent, and performing the study will be done in the private single oom, will only be reported in aggregate, not by individuals. No data will be linked to any information that could identify the subject To Participants It o Participants It all categories of costs that participants or their insurance companies will be responsible for: Participants will have no costs associated with this study Study related procedures that would be done under standard of care Study related procedures not associated with standard of care |

#### 2. If Other, explain: 3. \* Provide details of all financial costs to the participant, other than time and transportation. Additional details regarding

4. If applicable, upload a Cost Analysis form here:

ID: HM20005575

View: SF - Compensation

# Compensation

- 1. \* Describe any compensation that will be provided including: items such as parking/transportation
- total monetary amount
- type (e.g., gift card, cash, check, merchandise, drawing, extra class credit)
   how it will be disbursed:

standard of care costs will be requested on another screen, if applicable

2. If compensation will be pro-rated, explain the payment schedule:

ID: HM20005575

View: SF - Risks, Discomforts, Potential Harms and Benefits

# Risks, Discomforts, Potential Harms and Benefits

- 1. \* Describe the risks to participants associated with this study:
- physical, psychological, social, legal, financial, and other risks
- probability or likelihood of given risks
- 1. For some participants, the nasograstric tube may need to be replaced before the study begins. There is very very small risk of trauma, bleeding or a transient drop in heart rate when a new tube is placed. Note that tubes are placed and replaced routinely in this population. 2. Even though both modes of non-invasive ventilation are currently used clinically, it is possible that one mode will not be as well tolerated as the other, or that it will take longer than one hour to adjust the settings. The subject might have more apnea/bradycardia/desaturation events. While these are common and are, in fact, why the patient is being treated clinically with one of the two modes under investigation, a significant increase in the events. If this occurs, the study will be stopped and the clinical team notified. Any needed interventions will be under the direction of the clinical team. The most likely outcome will be to place the subject back on the ventilation mode that he/she was on prior to the study.

  3. The adverse events are the outcomes that will be affected by/measured for the interventions. Both NIPPV and NAVA are used to
- treat/prevent these events. The study is seeking to answer which mode is better at preventing them. Since we don't know this yet, it is possible that one of the modes will be worse, which is why it will be monitored as an adverse event, and if one mode does cause more events, the study will be stopped. Plus this info will be given to the clinician to use when selecting a mode for the patient in the future.
- 2. \* Describe how the risks / harms will be minimized:
- The nasogastric tubes will be placed by experienced NICU personnel who place nasogastric tube every day.
   The subjects will be monitored continuously by: cardiorespiratory monitor, 2 pulse oximeters and by direct observation by study personnel during the set-up phase and each four hour observations. If , during the first trial, the event number or severity increases beyond what which would be considered safe in normal clinical care, the mode will be considered a failure. The clinical team will be informed and the clinical team (not the investigators) will decide if, in their judgment, the alternate mode should be used for the second trial. If the increased event number or severity occurs during the second trial, the mode will be considered a failure, the clinical team will be informed and the clinical team will determine further care decisions.
- 3. The events are ones that are monitored as part of the usual care, and this will continue during the study period. These babies are always connected to monitors which are linked to nursing phones as well as central telemetry. The investigator doing the study will be present to assess/intervene, and as back-up, the clinical team will provide their routine care for such events
- 3. If the disclosure of any of the information obtained during the study would place the individual at risk for harm (legal, reputation, emotional etc.) and the information will be recorded so that the individual could be identified, explain the protections that will be put in place to decrease the risk of disclosure:
- 4. \* The Code of Virginia requires that most medical personnel and all employees of institutions of higher education report suspected child/elder abuse or neglect. Is it likely investigators could discover information that would require mandatory reporting by the investigators or staff:
- No
- 5. \* Is it likely investigators could discover a participant's previously unknown condition (eg disease, suicidal thoughts, wrong paternity) or if a participant is engaging in illegal activities:

  - No
- 6. If yes, explain how and when such a discovery will be handled:
- 7. \* Describe any potential risks or harms to a community or a specific population based on study findings: None anticipated
- 8. \* Describe criteria for withdrawing an individual participant from the study; such as safety or toxicity concerns, emotional distress, inability to comply with the protocol, etc.:
- If, between consent and study, the subject no longer meets inclusion criteria or does meet exclusion criteria If the number/severity of events becomes a clinically relevant safety concern, the study mode will be considered a failure. The clinical team will be informed and they will have the authority to stop the study.
- 9. \* Summarize any pre-specified criteria for stopping or changing the study protocol due to safety concerns:
- The exact number/severity of events that might define a safety concern is subject dependent based on prior event history. A subject who normally has 0-1 events an hour may have a clinical safety concern at 4-5 events/hr while in one who is normally having 3-4 events/hr, the same rate of 4-5 events would not be significant. Clinically, a change in event rate is judged against baseline rate. However, events that require significant intervention, i.e. mechanical breathing support from ventilator or bag and mask, will be an absolute stopping
- The threshold for an adverse event will be dependent on the baseline level. If the baseline rate is, say, 4-6 events an hour, a 25% increase is 1 event, which is within the patient's variance. On the other hand, in one having no events, just one event is a 100% increase. We have 2 criteria - 1) An event that requires intervention with breathing support such as with more breaths or a bag and mask, 2) an increase from baseline of at least 4-5 events/hr, from baseline
- 10. Where appropriate, discuss provisions for ensuring necessary medical, professional, or psychological intervention in the event of adverse events to the subjects: Current protocols in place in NICU.
- 11. \* Describe any potential for direct benefits to participants in this study: Observational results will be shared with the clinical team. These may include infant's comfort level on each mode of non-invasive ventilation; pressure levels on each mode, general frequency of apnea/bradycardia/desaturation events. Based on this information, the clinical team may choose to change the mode of ventilation.
  - There are no well-characterized tools to measure premature infant 'comfort'. There are semi-subjective pain scores that the nursing staff use but we are more likely to have irritation or discomfort from the probe. Thus, this will be an ongoing assessment of a) the infant's state - quiet sleep, quiet awake, agitated, restless, etc. b) new onset tachycardia or tachypnea coincident with applying the probes. c) facial grimaces that are different than baseline as assessed by the nurse caring for the patient.
- 12. \* Describe the scientific benefit or importance of the knowledge to be gained:

Information derived from analysis of study data may determine which mode of non-invasive ventilation is better in short term use for VLBW infants by examining outcome data with more depth and precision than is currently done clinically. This will help clinicians to better choose the optimal mode.

13. If applicable, describe alternatives (research or non-research) that are available to potential participants if they choose not to participate in this study:
They will be maintained on their current clinically chosen mode of ventilation 14. \* Indicate if this study will have a Data Safety Monitoring Board (DSMB) or a Data Safety Monitoring Plan (DSMP): [Required for all Full Review studies] DSMB Review Required DSMP Required Not Required ID: HM20005575 View: SF - DSMP Details

# DSMP Details

1. \* Describe your Data Safety Monitoring Plan for monitoring the data collected to ensure the safety of participants: At 5 subject intervals, data on the number of failures, and the frequency/severity of events will be provided to Dr. Karen Hendricks-Munoz, MD, MPH who is Chair of Neonatal Medicine at VCU. She will assess the study for safety. Her opinion about whether the study should continue is final.

The DMSP is the chief of the service. We will submit outcomes and adverse event data to her after every 5 subjects. It is an expectation that the DMSP assessment of whether to stop or continue will be made in writing to the PI within 28 days, and a copy will be forwarded to the other investigators, the device sponsor and the IRB each time.

ID: HM20005575

View: SF - Consent Qualifiers

# Consent Qualifiers

1. \* Are you submitting your study as exempt and therefore no consent is required:  $\hfill \hfill \$ 

No

ID: HM20005575

View: SF - Consent Groups

# Consent Groups

1. \* List all consent groups:

| Group | Types | Waivers | Roles | - | Consent | Coercion | Decision | Status<br>Change |
|---|---|---|---|---|---|---|---|---|
| | | | | Other | | | | |
| VLBW<br>infants on<br>non-<br>invasive<br>ventilation | Parent/Guardian | No<br>Waivers<br>Requested | Principal<br>Investigator<br>Co/Sub-<br>Investigator<br>Trainee/Student | t | In the subject's private room when the parents/guardians are visiting | Preference will be given to having one of the investigators not currently caring for the potential subject as person to obtain consent. The alternative of not participating, with no effect on care, will be emphasized during review of the consent form Several of the investigators take one week turns on the clinical service where the study participants will be cared for. Since only the investigators will be obtaining consent, it is very likely that an investigator who is not directly caring for the patient will be available to explain the study and obtain consent. Since the subjects are usually in the NICU for weeks, during which they often meet the criteria to participate, it would be very unusual for the clinician caring for the subject to need to get consent | invasive<br>ventilation | |

2. Upload any consent / assent documents:

View: SF - Documents ID: HM20005575

# Documents ID: HM20005575 View: SF - Protocol Complete Section Complete: SUMMARY End of Application: IRB HUMAN SUBJECTS STUDY Click Continue Below



| o-Med Devices |
|-------------------------------|
| new use of a marketed device: |
| r the device: |

- VCU Sponsor who is not the Investigator
- Not Required
- 5. If evaluating an approved device, upload documentation of the approved uses:  $\mbox{Servo-i}\ (0.01)$

Describe use of the device in the methods section.

ID: HM20005575

View: Bio-Med Devices

# **Bio-Medical Devices**

1. \* Name: Servo-i NAVA

2. \* Manufacturer: Maquet

- 3. \* Provide the IDE number for any investigational devices or new use of a marketed device:  $\ensuremath{\text{N/A}}$
- 4.  $^{\star}$  Select who holds the Investigational Device Exemption for the device:

| External to VCU Sponsor or Investigator |
|-----------------------------------------|
| VCU Sponsor-Investigator |
| VCU Sponsor who is not the Investigator |
| Not Required |

# 5. If evaluating an approved device, upload documentation of the approved uses: NAVA brochure (0.01) $\,$

Describe use of the device in the methods section.